CLINICAL TRIAL: NCT07104656
Title: Evaluate How Use of an Inferior Border Saw While Making the Inferior Border Osteotomy During Sagittal Ramus Osteotomy Using the Low and Short Medial Osteotomy Modification Technique Affects the Lingual Fracture Pattern of the Mandible
Brief Title: Bony Overlap Following Use of the Inferior Border Saw for the 'Low and Short' Sagittal Split: A Split-Mouth Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Brian Kinard, Principal Investigator, University of Alabama at Birmingham
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-300014869; UAB (Other: UAB)
Record Dates: First submitted 2025-07-29; First posted 2025-08-05 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Mandibular Surgery
Keywords: Mandibular; osteotomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Participants receiving right jaw surgery (Active Comparator): Participants receiving inferior border saw on right jaw surgery
  Interventions: Procedure: Inferior Osteotomy made by border saw; Procedure: Inferior Osteotomy made with reciprocating saw
- Participants receiving left jaw surgery (Active Comparator): Participants receiving inferior border saw on left jaw surgery
  Interventions: Procedure: Inferior Osteotomy made by border saw; Procedure: Inferior Osteotomy made with reciprocating saw

INTERVENTIONS:
Procedure: Inferior Osteotomy made by border saw — Inferior border saw used to make the inferior border osteotomy
Procedure: Inferior Osteotomy made with reciprocating saw — reciprocating saw used to make the inferior osteotomy

SUMMARY:
The purpose of this study is to evaluate if use of an inferior border saw while making the inferior border osteotomy is associated with the medial cortex fracture pattern.

ELIGIBILITY:
Inclusion Criteria:

* patient's having mandible surgery

Exclusion Criteria:

* Severe dentofacial deformity secondary to a syndromic diagnosis

Ages: 12 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-01-07 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Type Medial Cortex Fracture Pattern | 5 weeks
  CT scan comparison of the lingual cortex of the mandible to evaluate the fracture pattern. Classified into 4 fracture patterns (Using the Lingual Split Scale.) On a scale of LSS1 vertical Fracture, LSS2 Horizontal Fracture, LSS3 Fracture along the mandibular canal, LSS4 unfavorable fracture. Where 1, 2, and 3 are favorable and 4 is unfavorable.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: Undecided